CLINICAL TRIAL: NCT04296370
Title: A Phase III, Open Label, Randomised, Controlled, Multi-centre Study to Assess the Efficacy and Safety of Fluzoparib±Apatinib Versus Physicians Choice Chemotherapy in the Treatment of HER2-negative Metastatic Breast Cancer Patients With Germline BRCA1/2 Mutations
Brief Title: A Study of Fluzoparib±Apatinib Versus Chemotherapy Treatment of Physician's Choice in HER2-negative Metastatic Breast Cancer Patients With Germline BRCA Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-Ⅲ-303
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-03

CONDITIONS: Treatment in HER2-negative Metastatic Breast Cancer Patients With Germline BRCA Mutation
MeSH Terms: interventions — fluzoparib; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety Lead-in, Doublet Arm (Experimental): Fluzoparib+Apatinib
  Interventions: Drug: Fluzoparib; Apatinib
- Single Arm (Experimental): Fluzoparib
  Interventions: Drug: Fluzoparib
- Physician's choice chemotherapy (Active Comparator): Capecitabine or Vinorelbine
  Interventions: Drug: Physician's choice chemotherapy

INTERVENTIONS:
Drug: Fluzoparib; Apatinib — Fluzoparib Orally twice daily; Apatinib Orally once daily
  Arms: Safety Lead-in, Doublet Arm
Drug: Fluzoparib — Fluzoparib Orally twice daily
  Arms: Single Arm
Drug: Physician's choice chemotherapy — Investigators will declare one of the following regimens:
  Capecitabine Vinorelbine
  Arms: Physician's choice chemotherapy

SUMMARY:
This is a multicenter, randomized, open-label, 3-arm Phase 3 study to evaluate the efficacy and safety of Fluzoparib alone or with Apatinib versus Physicians Choice Chemotherapy, as treatment, in patients with a Germline BRCA Mutation and HER2-negative Metastatic Breast Cancer. The study contains a Safety Lead-in Phase in which the safety and tolerability of Fluzoparib+Apatinib will be assessed prior to the Phase 3 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* （Saftey Lead-in + phase 3）Germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious
* （Saftey Lead-in + phase 3）human epidermal growth factor receptor type 2 (HER2)-negative metastatic breast cancer
* （Saftey Lead-in + phase 3）had received ≤2 lines of chemotherapy for mBC
* （Saftey Lead-in + phase 3）Prior therapy with an anthracycline and a taxane in either an adjuvant or metastatic setting.
* ER/PR breast cancer positive patients must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy.
* ECOG performance status 0-1.
* Adequate bone marrow, kidney and liver function.

Exclusion Criteria:

* Prior treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor or Apatinib
* Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry. Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix, DCIS or stage I grade 1 endometrial cancer allowed
* Radiation or anti-hormonal therapy or other targeted anticancer therapy within 14 days before randomization
* Known to be human immunodeficiency virus positive
* Known active hepatitis C virus, or known active hepatitis B virus
* Untreated and/or uncontrolled brain metastases
* Pregnant or breast-feeding women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
(Safety Lead-in) dose limited toxicity (DLT) | up to 21 days
  dose limited toxicity (DLT) of Fluzoparib+Apatinib in the first cycle
(Safety Lead-in) Recommended Phase II Dose (RP2D) | up to 21 days
  Recommended Phase II Dose (RP2D) of Fluzoparib+Apatinib
(Phase 3) Progression free survival(PFS) in HER2-negative Metastatic Breast Cancer patients | Radiological scans performed at baseline then every ~6 weeks up to 30 weeks, then every ~ 9 weeks thereafter until objective radiological disease progression. Assessed up to a maximum of 30 months
  Defined as progression free survival per RECIST 1.1 criteria according to BIRC criteria

SECONDARY OUTCOMES:
AEs+SAEs | from the first drug administration to within 30 days for the last treatment dose
  Adverse Events and Serious Adverse Events
PFS by investigator's assessment | up to 30 months
  Progression-Free-Survival
OS | up to 30 months
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up
Patient Reported Outcomes (PROs) assessed by EORTC QLQ C30 questionnaire | up to 30 months
  Comparison of the Quality of Life in study arms assessed by EORTC QLQ C30 questionnaire
Time to progression on the next anticancer therapy (PFS2) | up to 30 months
  From date of start of next anticancer therapy to date of first documented progression of date of death from any cause, whichever comes first
Objective Response Rate (ORR) | up to 30 months
  Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by CT or MRI
Disease control rate (DCR) | up to 30 months
  Complete response + Partial response + Stable disease (CR+PR+SD) based on RECIST 1.1
Duration of response (DoR) | up to 30 months
  Time from documentation of tumor response to disease progression assessed among patients who had an objective response

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu HengRui Medicine Co., Ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Liu J, Ouyang Q, Wang S, Liu Y, Teng Y, Wang X, Cheng J, Tong Z, Sun T, Yan M, Zhou X, Li F, Nie J, Shao ZM, Ye C, Wang Y, Wu X, Li Z, Wu Y, Xiong H, Li H, Gan L, Niu Z, Zhang J, Zhang Q, Pan Y, Wu X, Zhang Y, Xie W, Xiao Y, Gao J, Zhao H, Yin Y, Qian Z, Sun S, Zhang H, Wang K, Lu J, Li Y, Wang X, Yang X, Wang Y, Wang Q, Song E. Fuzuloparib with or without apatinib in patients with HER2-negative metastatic breast cancer with germline BRCA1/2 mutations (FABULOUS): interim analysis of a multicentre, three-arm, open-label, randomised, phase 3 trial. Lancet Oncol. 2025 Dec;26(12):1563-1574. doi: 10.1016/S1470-2045(25)00523-6. PMID 41308673